CLINICAL TRIAL: NCT05689814
Title: A Single-centre, Randomised, 3-way Cross-over, Clinical Investigation Comparing Denture Fixative Versus no Fixative Performance in Full Denture Wearers and an Exploratory Substudy in Partial Denture Wearers
Brief Title: Retention, Stability and Performance Assessment of Denture Fixatives Versus no Fixative Control
Acronym: RESONATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Reckitt Benckiser Healthcare (UK) Limited (Industry)
Collaborators: University of Leeds (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 0708501
Record Dates: First submitted 2022-12-09; First posted 2023-01-19 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Dentures
Keywords: Denture Fixative

STUDY DESIGN:
Intervention Model Description: The denture fixative cream formulations will be tested in a 3-arm cross-over-design, where subjects will be randomised to a sequence including the two intervention (denture fixative) arms and a control (no fixative) arm.
Who Masked: Outcomes Assessor
Masking Description: Masking versus no fixative control will not be possible, however, clinical outcomes assessors will be masked to the two different investigational denture fixative products
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Paraffin based Denture Fixative (Experimental): Participants will use the paraffin-based denture fixative to secure their denture for 4 days and an additional 21-35 days during the observational (safety) period in accordance with the randomization schedule.
  Interventions: Device: Paraffin based Denture Fixative
- Polydecene based Denture Fixative (Active Comparator): Participants will use the polydecene based denture fixative to secure their denture for 4 days and an additional 21-35 days during the observational (safety) period in accordance with the randomization schedule.
  Interventions: Device: Paraffin based Denture Fixative
- No Denture Fixative Control (No Intervention): Participants will continue to wear their dentures for 4 days and will not use any denture fixative as part of this study arm.

INTERVENTIONS:
Device: Paraffin based Denture Fixative — Denture fixative applied in strips to secure dentures in place
  Other Names: Denture Fixative
  Arms: Paraffin based Denture Fixative; Polydecene based Denture Fixative

SUMMARY:
This clinical investigation will evaluate the effectiveness, tolerability and safety of two denture fixative creams versus no fixative control

DETAILED DESCRIPTION:
A single-centre, randomised, 3-way cross-over, clinical investigation comparing the performance of two denture fixative versus no denture fixative control in full denture wearers and an exploratory sub study in partial denture wearers. The study will assess the performance and tolerance of two denture fixative cream formulations (Paraffin based and Polydecene based) when applied to full dentures.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with a completely edentulous maxillary [UPPER] arch restored with a conventional full acrylic-based complete denture and dentate, partial, or full edentulous mandibular [LOWER], which may be restored with a stable complete, partial or implant supported denture
2. For complete denture wearers, maxillary [UPPER] dentures must be completely removable standard acrylic dentures, which are at least moderately well-fitting at the screening visit (modified (Olshan) Kapur Index: retention score ≥2, stability score ≥2)
3. Male or female participants aged between 18 and 85 years at the time of signing the informed consent form
4. Participants must have been using dentures daily for at least 6 months prior to the screening visit
5. Dentures must have been made in the last 5 years;
6. Dentures must be well-made based on design and construction in the opinion of the clinician
7. No clinically significant and relevant abnormalities in medical history or upon oral examination

Exclusion Criteria:

1. Female participants who are pregnant as confirmed by a positive pregnancy test (urine) or are lactating (applicable to female participants of childbearing potential)
2. Daily doses of medication that might interfere with the ability to perform the study according to protocol or affect study assessments, for example, bisphosphonates (oral or intravenous) (as determined by the Investigator)
3. Known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients
4. Any clinically significant or relevant oral abnormality (e.g., temporomandibular joint [TMJ] problems), or recent (within last 6 months) oral surgery / intervention, or oral health concern that, in the opinion of the investigator, could affect the participant's participation in the study
5. Participants with maxillofacial defects covered by prosthetics
6. Self-reported and/or visual manifestations of severe dry mouth (xerostomia) that may affect denture retention in the opinion of the Investigator
7. Participants with oral soft tissue examination findings such as stomatitis, open sores, ulcers, lesions, redness or swelling or associated lymphadenopathy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2023-01-30 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Denture Retention Assessment at 1hour | 1 hour after denture fixative application or no fixative control
  To assess denture retention of full maxillary arch after 1 hour with and without denture fixative using the Modified (Olshan) Kapur Index. Retention will be measured on score of 0-5 to assess the nature of resistance offered by the denture/denture fixative to vertical force. The higher the score, the higher the retention ability of the denture and fixative.

SECONDARY OUTCOMES:
Denture Retention Assessment at 5minutes and 30minutes | 5mins and 30 mins after denture fixative application or no fixative control
  To assess denture retention in full maxillary arch (and mandibular arch in fully edentulous participants) using the Modified (Olshan) Kapur Index at 5 and 30 minutes. Retention will be measured on score of 0-5 to assess the nature of resistance offered by the denture/denture fixative to vertical force. The higher the score, the higher the retention ability of the denture and fixative.
Denture Stability at 5minutes, 30minutes and 1hour | 5mins and 30 mins after denture fixative application or no fixative control
  To assess denture stability in full mandibular arch (if present) using the Modified (Olshan) Kapur Index as separate scores at 5minutes, 30 minutes and 1 hour.
Denture Hold Assessment | ≤2 hours, 2 to 4 hours, 4 to 6 hours and 6 to 12 hours after denture fixative application or no fixative control
  To assess denture hold (retention and stability) at ≤2 hours, 2 to 4 hours, 4 to 6 hours and 6 to 12 hours using the Modified (Kulak) Kelsey questionnaire compared to no fixative control
Gum Comfort Assessment | At the end of each participant's day during the 4-day treatment period for each arm
  To assess gum comfort using the Gum Comfort questionnaire comparing denture fixative to no fixative control over periods of 4 days (change in overall mean score and individual responses)
Participant Satisfaction Assessment | At the end of each participant's day during the 4-day treatment period for each arm
  To assess participant satisfaction of the denture fixatives using the Modified (Kulak) Kelsey questionnaire compared to no fixative control
Oral Health Assessment | To be completed once during the participant's clinic visit on days 2,3,4,5,6,7 and 8 comparing with and without fixative
  To make a clinical assessment of the oral health impact profile of participants using the Oral Health Impact Profile-Edentulous (OHIP-EDENT) questionnaires after 4 days use of each of the dental fixatives administered and no fixative control.
Bite Force Assessment | To be completed once during the participant's clinic visit on days 3, 5 and 7
  To measure Bite force by means of a digital gnathometer to compare the denture fixatives to no fixative control

CONTACTS AND LOCATIONS:
Overall Officials: Sue Pavitt, Professor, Principal Investigator — Dental Translational and Clinical Research Unit, School of Dentistry, University of Leeds, UK
Locations (1):
- Dental Translational and Clinical Research Unit, School of Dentistry, University of Leeds, Leeds, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
IPD will be shared if required as per local regulations